CLINICAL TRIAL: NCT05847075
Title: Effect of Heat Therapy Compared With Strength Training on Metabolic Profile, Heat Shock Response, Inflammation, Cardiovascular Responses and Microbiota in Individuals With Type 2 Diabetes
Brief Title: Heat Therapy and Strength Training Effects in Individuals With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Maurício Krause, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38626420.6.0000.5347
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
Keywords: Heat Therapy; Inflammation; Metabolism; Microbiota; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperthermia; Inflammation; Diabetes Mellitus | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Volunteers who meet the inclusion criteria will be guided in the study and asked to sign a written informed consent before enrollment in the trial. Participants will be randomized into intervention groups Control (C), Resitance/Strength training (RT) or Heat Therapy (HT).
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, the researcher conducting the exercise sessions as well as participants will not be blinded. To ensure assessor masking, the subjects are asked to omit their assigned group and not to talk about their interventions during the outcome evaluation sessions. In the case of unintentional unblinding for any reason, the involved researcher will notify the principal researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary Diabetic people (Experimental): Sedentary people with Type 2 Diabetes.
  Interventions: Other: Sedentary Control
- Heat Therapy (Experimental): Diabetic people allocated in Heat Therapy for 12 weeks.
  Interventions: Other: Heat Therapy
- StrengthTraining (Experimental): Diabetic people allocated in Strength training for 12 weeks.
  Interventions: Other: StrengthTraining

INTERVENTIONS:
Other: Heat Therapy — Participants in the HT group will undertake whole body heat treatment according to previous methods. Participants will be housed in an environmental chamber initially set at 55.0oC on three non-consecutive days of the week during 12 weeks. Each session will last 60 min.
  Arms: Heat Therapy
Other: StrengthTraining — Participants will perform supervised exercise in a gym on three non-consecutive days of the week. Each session will last ~60 min and will consist of a warm up, the resistance training and a cool down. All sessions will be conducted by qualified sport and exercise scientists for 12 weeks.
  Arms: StrengthTraining
Other: Sedentary Control — Participants will not receive any intervention during 12 weeks.
  Arms: Sedentary Diabetic people

SUMMARY:
The aim of this study is to compare different non-pharmacological interventions in Type 2 diabetic people, testing their efficiency to improve metabolism and inflammation. The investigators will compare the effects of Heat Therapy (HT) and Strength training (ST), for 12 weeks, to test which one is more effective to improve participants health. Heat Therapy consists in submitting a person to an environmental chamber, initially set at 55 degrees Celsius on three non-consecutive days of the week. Each session will last 60 min. ST consists in supervised exercise in a gym on three non-consecutive days of the week. Each session will last ~60 min and will consist of a warm up, the resistance training and a cool down. All sessions will be conducted by qualified sport and exercise scientists for 12 weeks. A third group of people will stay sedentary without any other intervention for 12 weeks. Before, and after the end of the intervention blood samples will be collected to analyze metabolic parameters as well as inflammatory markers. The investigators hypothesize that ST and HT will reduce HbA1c levels, improve metabolic and inflammatory profile, dysbiosis, and the anti-inflammatory heat shock response (HSR).

DETAILED DESCRIPTION:
Materials and Methods Study design and setting The study is a prospective, randomized, double-blind, parallel, non-inferiority clinical trial, and will be conducted at Universidade Federal do Rio Grande do Sul, a University in Southern Brazil. This study protocol adheres to the SPIRIT recommendation.

Interventions Volunteers who meet the inclusion criteria will be guided in the study and asked to sign a written informed consent before enrollment in the trial. Participants will be randomized into intervention groups Control (C), RT or HT. In the control group, participants will not receive any intervention. In the intervention group RT, participants will perform supervised exercise in a gym on three non-consecutive days of the week. Each session will last ~60 min and will consist of a warm up, the resistance training and a cool down. All sessions will be conducted by qualified sport and exercise scientists for 12 weeks.

RT program will consist of a combination of upper and lower body exercises using gym equipments, free weights and body weight (functional exercises) as the primary resistance. The 12 weeks RT will be divided into three mesocycles of four weeks each (please see details of sets, repetitions and intervals in Table 1). Exercises will include leg press, knee extensions and leg curls, biceps curls, triceps extensions, lat pull down, shoulder press, bench press and abdominal crunch. Before the start of the training period, subjects will complete a familiarization session to practice the exercises they would further perform during the training program, when the exercise load was individually tested. The resistance training will be performed using two to three sets per exercise at intensities between 12 and 15 maximum repetitions (the heaviest possible weight to perform a total of 12-15 repetitions). The intensity of the functional exercises was controlled by OMNI scale. Each session will last 60 min.

Participants in the HT group will undertake whole body heat treatment according to previous methods. Participants will be housed in an environmental chamber initially set at 55.0oC on three non-consecutive days of the week. Each session will last 60 min. During the sessions, rectal temperature, heart rate, blood pressure and heat discomfort will be constantly measured.

Strategies for trial retention Participants will be asked once a week on the face-to-face visit to monitor their adverse events. Moreover, phone calls or messages will also be used to remember participants regarding scheduled or missed visits.

Recruitment and participant timeline The recruitment period for the study will be from April 2023 to December 2025. Participants will be invited to participate in the study by announcement in newspaper, electronic and social media. Figure 1 shows the flowchart of the study design.

Adherence Adherence to an exercise program has been classified as meeting at least 80% of the recommended or prescribe exercise dose. Any participant who demonstrates a training protocol adherence of 80% or more than 36 sessions will be considered adherent. Participants will be classified as non-adherent or partially adherent if their adherence is less than 80%.

Statistical considerations For assessment of exercise effect on Plasma HSP levels between groups post intervention, we assumed an 80% power, a 5% significance level, and a effect size (Cohen's F) of 0.4. We estimated a 10% dropout rate and the total number calculated was 22 in each group.

The randomly assigned participant's data will be analyzed according to the intention-to-treat principle as primary choice and to the per-protocol principle, with treatment, time and treatment-time interaction registered as the fixed effects. We will qualitatively document reasons and details of each case of withdrawal. The normality of the data will be tested by the Shapiro-Wilk test. Mean and standard deviation will be used to describe the parametric continuous variables and the median and interquartile range for non-parametric variables, while absolute and relative frequencies will be used for categorical variables. Analysis of variance (ANOVA) will be used to compare the final values of outcomes. Treatment effects (group, time, and group interaction) will be estimated using Generalized Estimation Equations (GEE) followed by the Bonferroni posthoc test (P < 0.05). A multiple linear regression analysis (backward method) will be performed to investigate the impact of routine pharmacotherapy, sex and age on the primary and secondary outcomes. The Statistical Package for Social Science Professional software version 20.0 (IBM Corp., Armonk, NY, USA) will be used for these analyses.

Allocation Participants will be randomly assigned to the groups according to a sequence of computer-generated random numbers. This sequence will be obtained in the Excel Microsoft program, in a 1:1 ratio, with blocks of eight or six participants to complete the total number calculated. A sealed envelope containing the allocation code will be opened only at the beginning of treatment in the participant's presence, according to the order of entry into the study.

Due to the nature of the interventions, the researcher conducting the exercise sessions as well as participants will not be blinded. To ensure assessor masking, the subjects are asked to omit their assigned group and not to talk about their interventions during the outcome evaluation sessions. In the case of unintentional unblinding for any reason, the involved researcher will notify the principal researcher.

Data collection and management A questionnaire will be applied to obtain the sociodemographic and clinical characteristics of participants, including age, sex, marital status, schooling level, diabetes duration, family history of diabetes, and self-reported physical activity. Drugs for T2DM will be registered at baseline and the end of the study.

Anthropometry measures, including body weight, height, calculated body mass index (kg/m2), waist, and hip circumferences changes, will be recorded at the first and last visit. The weight will be measured in a digitally calibrated balance with a maximum capacity of 150 kg and a precision of 100 g. The height will be determined by a vertical stadiometer attached to the balance with a capacity of 2 m/0.1 cm (Urano®, Canoas, Brazil). Waist and hip circumferences will be measured with an inelastic metric tape (2 m/0.1cm). Total corporal composition will be evaluated through dual-energy X-ray absorptiometry (DEXA scan - Lunar iDXA, GE Healthcare, Buckinghamshire, UK).

After this evaluation, individuals will perform a self-limited maximal exercise test on a treadmill to determine peak oxygen uptake (VO2 peak) and peak heart rate, supervised by a team of experienced exercise physiologists. The test will be carried according Bruce protocol. Oxygen uptake (VO2) and carbon dioxide production (VCO2) will be determined by a breath-by-breath computerized gas exchange system and analyzed using at a 20-second averaging signal. Basal metabolic rate will be analyzed in fast state (Quark CPET, Cosmed, Italy).

At the first and last visit to the laboratory, blood samples will be collected and centrifuged at 1000 g for 10 minutes to separate plasma or serum, which will be stored for further analysis of biochemical parameters. Total glucose, C-reactive protein, HDL-cholesterol, HbA1c, and triglycerides will be determined in an automated system Cobas C111 (Roche Diagnostics, Basel, Switzerland). LDL-cholesterol will by calculated by the Friedewald equation. Insulin resistance will be calculated by the Homeostatic Model Assessment (HOMA-IR) method, based on insulin and fasting glucose levels.

To microbiota analysis, silica-membrane-based DNA purification from feces will be performed by the high quality nucleic acid extraction commercial kit QIAmp Blood and Body Fluid (Qiagen, Canada). The V3-V4 hypervariable region of the 16 S rRNA gene will be amplified and sequenced on an Illumina MiSeq. Sequences will be processed in mothur (v.1.41.1) 23 with modified procedures, as previously described. Sequences will be then aligned to the SILVA 16 S rRNA database (v 132).

For inflammatory biomarkers and plasma LPS levels, the blood will be centrifuged at 1000 g for 10 minutes and serum will be frozen (-80 °C) for further analysis by the enzyme-linked immunosorbent assay (ELISA) technique, using commercial kits: LPS, TNF-α, IL-1, IL-4, IL-5, IL-6, IL-10, and IL-13 (Human ELISA Kits, Sigma-Aldrich, St. Louis, MI, USA).

Considering the importance of the HSR for stress adaptation, we will test the capacity of leukocytes (a major source of circulating HSP72 and representative of immune cell stress response), to release HSP72, under heat stress conditions (a normal and expected response in healthy cells). We will use this strategy to compare if different intervention could improve the HSR in diabetes. Briefly, after harvesting, whole blood was immediately incubated at two different temperatures: 37 °C (control) and 42 °C (heat stressed) for 2 h in a water bath. After incubation, total blood will be centrifuged to isolate plasma. Plasma will be used for the analysis of eHSP72 26. A highly sensitive, enzyme-linked immunosorbent assay (EIA) method (EKS-715 Stressgen, Victoria, Canada) will be used to quantify the levels of plasma HSP72 protein as previously described 27. Inflammatory cell signaling in PBMC (NF-kB; TLR2 e 4, TRIF, IKKi/IKKε, e MyD88) will be analyzed by western blot, as previously described 28.

Flow mediated dilation Brachial artery flow mediated dilation (FMD), in response to hyperemia, will be performed using an ultrasound device (Toshiba model Nemio XG, Japan) as an indirect measurement of endothelial function, adapted to current guidelines . (THIJSSEN DHJ et.al., 2011).

Hydration protocol On the previous day of heat exposure, participants will be instructed to drink 12 mL•kg-1 of water (in addition to the usual liquid consumption). During the morning of the day of the experimental session in the heat, the participants will be instructed to consume 6 mL•kg-1 of water, in addition to the usual liquid consumption, to ensure the state of euhydration. Prior to entering in the environmental chamber, a urine collection will be performed to verify the state of hydration, using the specific gravity through a refractometer 29; 30 and the color through a specific scale 31. A urine specific gravity cutoff of 1.25 will be applied. For higher values, participants will drink 200-250 mL of water and wait 30 minutes before the heat exposure.

Safety and adverse events Participants will be under continuous health professional control during and at least 30 min after the intervention to prevent adverse events. The following mild and moderate adverse events can appear: Exercise protocols, particularly during maximum effort, can cause some discomfort (nausea, muscle soreness). Heat therapy has been shown to be safe for most people. However, for some participants, it is possible that the higher temperature causes some thermal discomfort. The cardiovascular changes, such as increased heart rate and blood pressure, are expected and not harmful. Finally, a mild dehydration may be observed after the protocol. This will be attenuated with proper hydration afterwards.

Ethical Considerations The study strictly follows the protocols regarding informed consent form, confidentiality, and anonymity. An informed consent form with guidelines, objectives of the project, description of procedures, possible risks, and benefits will be provided. Participants will be also informed that participation is voluntary, and they can withdraw from the study at any time. This study will be conducted in accordance with the Declaration of Helsinki and was approved by the facility's institutional review board (Tracking number: 38626420.6.0000.5347) and registered in the Clinical Trials Database. All files containing the participants' data will be stored in a secure database password-protected document that will be accessed only by authorized members of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* HbA1c levels were between 7.0% and 10%
* Sedentary
* Non-smoking
* Body mass index (BMI) between 18.5-39.9 kg/m2,
* No use of insulin.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Under treatment with antibiotics or anti-inflammatory drugs within 4 weeks,
* History of cardiovascular diseases: myocardial infarction, cardiac illness, vascular disease, stroke, or any condition that would prevent them from engaging in an exercise study;
* Engaged in two or more planned and structured exercise sessions per week (in the last six months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Plasma HSP72 | First visit, prior to the intervention (baseline) AND 2 weeks of intervention.
  Plasma concentration (in ng/mL) of HSP72.

SECONDARY OUTCOMES:
Fasting glucose | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  Fasting glucose (mmol/L)
Insulin plasma concentration | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  Fasting Insulin (mlU/L)
Insulin resistance (HOMA-IR) | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  HOMA-IR (AU: arbitrary units)
Body Mass Index (kg·m-2) | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Visceral adipose tissue (VAT) | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  Visceral adipose tissue (mm): VAT measurements are performed with the subjects fasting, in supine position, and visceral fat is measured at the end of a normal expiration with the vertebral column positioned horizontally. VAT ultrasound measurements will be performed with a 38-mm, 3,75 -MHz convex-array probe that is placed directly above the umbilical scar. VAT thickness is considered as the distance between the posterior part of the rectus abdominal muscle and the posterior wall of abdominal artery.
Body composition | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  Dual-energy X-ray absorptiometry - DEXA scan - Measurements of total fat (%) and lean body mass (%).
Physical fitness (VO2 - Oxygen consumption) | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  VO2peak (mL O2/kg/min) - Oxygen uptake (VO2) and carbon dioxide production (VCO2) will be determined by a breath-by-breath computerized gas exchange system and analyzed using at a 20-second averaging signal (Quark CPET, Cosmed, Italy).
Gut microbiota DNA | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  To address the gut microbiota, the genomic DNA will be extracted from 0.25g of homogenized fecal samples using the QIAamp PowerFecal Pro DNA Kit (Qiagen, USA) according to manufacturer's instructions. Quality of the DNA will be evaluated by agarose gel electrophoresis and purity using 260/280 and 260/230 ratios measured by NanoDrop 1000 instrument (Thermo Fisher Scientific, Waltham, MA). DNA concentration will be quantified using Qubit dsDNA Reagent (Molecular Probes, Thermo Fisher Scientific division, Eugene, OR). The V3-V4 hypervariable region of the 16S rRNA gene will be amplified and sequenced on an Illumina MiSeq (2×300bp). The software package DADA2 will be used for taxonomic assignment (with SILVA database) and perform alpha and beta-diversity analysis in RStudio.
Inflammatory/anti-inflammatory markers | First visit, prior to the intervention (baseline) AND 12 weeks of intervention.
  Plasma concentration (in ng/mL) of C-reactive protein level, TNF, IL-1, IL-4, HSP72, IL-6, IL-10, adiponectin and leptin.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Krause, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Universidade Federal do Rio Grande do Sul, Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bock PM, Kowalewski LS, Ayres LR, Russo MKB, Leites GT, Martins AF, Oliveira AR, Krause M. Effect of heat therapy compared with strength training on metabolic profile, heat shock response, inflammation, cardiovascular responses and microbiota in individuals with type 2 diabetes: study protocol of a randomized trial. Sao Paulo Med J. 2025 Jun 2;143(3):e2024040. doi: 10.1590/1516-3180-2024.0040.R1.13082024. eCollection 2025. PMID 40465937